CLINICAL TRIAL: NCT06012760
Title: Effect of Iron Sucrose Combined With Human Erythropoietin and Vitamin C on Perioperative Allogeneic Red Blood Cell Infusion in Major Cardiac Surgery
Brief Title: The Effect of Combined Iron Protocols on Perioperative Allogeneic Transfusion
Acronym: CIPAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); The Central Hospital of Lishui City (Other); First Affiliated Hospital of Chongqing Medical University (Other); Zhejiang Provincial People's Hospital (Other); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); Zhejiang University (Other); Nanjing Hospital affiliated hospital of Nanjing medicine University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A2023519
Record Dates: First submitted 2023-08-22; First posted 2023-08-25 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-01

CONDITIONS: Anemia; Iron Deficiency Anemia; Perioperative; Transfusion; Cardiac Surgery
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — Ferric Oxide, Saccharated; Ascorbic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Iron Protocols group（CIP group） (Experimental): Preoperative randomization was conducted, followed by a three-day regimen in the week preceding surgery, involving the administration of intravenous iron sucrose at a dosage of 200 mg per day, vitamin C at a dosage of 2 g per day, and subcutaneous administration of Human Erythropoietin Injection at a dosage of 150 IU per kilogram.
  Interventions: Drug: Iron sucrose, Human Erythropoietin Injection, Vitamin C
- Standard Medical Care group（SMC group） (Active Comparator): Standard Medical Care (SMC) for the treatment of IDA. SMC as determined by the Investigator for the treatment of iron deficiency anemia (IDA).
  Interventions: Drug: Standard Medical Care

INTERVENTIONS:
Drug: Iron sucrose, Human Erythropoietin Injection, Vitamin C — The participants were administered a combined iron supplementation regimen consisting of iron sucrose,Human Erythropoietin Injection, and vitamin C, three times throughout the preoperative week.
  Arms: Combined Iron Protocols group（CIP group）
Drug: Standard Medical Care — Standard Medical Care (SMC) for the treatment of IDA. SMC as determined by the Investigator for the treatment of iron deficiency anemia (IDA).
  Arms: Standard Medical Care group（SMC group）

SUMMARY:
The goal of this clinical trial is to learn if a combined iron supplementation regimen can reduce the need for blood transfusions in adults with iron-deficiency anemia undergoing major elective cardiac surgery. The trial will also look at whether this regimen is safe and well tolerated. The main questions it aims to answer are:

Does the combined regimen lower the amount of allogeneic red blood cell transfusion needed during and after surgery?

Are there any side effects or safety concerns associated with the regimen?

Researchers will compare the combined iron supplementation (sucrose iron, erythropoietin, and vitamin C) to standard care to see if it helps reduce blood transfusions.

Participants will:

Receive either the combined regimen or standard care before surgery

Undergo major elective cardiac surgery under general anesthesia

Be monitored for blood transfusion needs and recovery up to 90 days after surgery

DETAILED DESCRIPTION:
1. Hypothesis:The combined protocol of preoperative sucrose iron, human erythropoietin, and vitamin C will demonstrate superiority in reducing perioperative allogeneic red blood cell (RBC) transfusion volume compared to standard care in patients with iron deficiency anemia undergoing major cardiac surgery with cardiopulmonary bypass.
2. Interventions 2.1.Experimental group: Patients in the experimental group will receive a combination therapy consisting of intravenous sucrose iron (200 mg), subcutaneous recombinant human erythropoietin (150 IU/kg), and intravenous vitamin C (2 g), administered once daily for three consecutive days within the week prior to surgery.

   2.2.Control group: Routine perioperative management based on clinical judgment, including observation, monitoring, and standard nursing practices.
3. Primary endpoint: Total volume of allogeneic RBC transfusion (units) from surgery initiation to postoperative day 5.
4. Stratification in randomization: Stratification factors include types of surgery, preoperative baseline hemoglobin level.
5. Follow-up time important points include: baseline upon hospital admission, the morning of surgery, postoperative day 1, postoperative day 5, at discharge, 30 ± 7 days after surgery, and 90 ± 7 days after surgery.
6. All perioperative transfusion decisions will follow standardized restrictive transfusion thresholds. When the patient's hemoglobin concentration falls below the threshold of 70 g/L during surgery or ICU monitoring, or below 70-80 g/L in the general ward, and/or when signs of anemia or hemodynamic instability are present-including shock, severe arrhythmias, respiratory distress, heart rate >120 beats/min, systolic blood pressure (SBP) <80 mmHg, mean arterial pressure (MAP) <55-60 mmHg, or a reduction in SBP or MAP exceeding 25% from baseline-these findings may indicate significant hypovolemia and warrant consideration of transfusion intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 18 years of age.
2. Major cardiac surgery should encompass procedures such as coronary artery bypass grafting (CABG), valve surgery, or a combination of both.
3. Iron deficiency anemia is defined as having a ferritin level below 100 μg/L or a ferritin level below 300 μg/L accompanied by a transferrin saturation below 25%. Additionally, hemoglobin levels should range between 90 and 130 g/L for men or between 90 and 120 g/L for women.
4. The American Society of Anesthesiologists (ASA) classification should fall within Grade 1-3.
5. Prior to participation, the patient or their legal representative must provide informed consent.

Exclusion Criteria:

1. Contraindications for the administration of iron sucrose, ascorbic acid, or rHuEPO.
2. Presence of a temperature exceeding 37.5 °C or the utilization of non-prophylactic antibiotics.
3. Individuals with a weight equal to or less than 50kg.
4. Individuals with a family history of haemochromatosis or thalassaemia, or those with a transferrin saturation level exceeding 50% or a documented history of iron overload.
5. Presence of other known haematological disorders such as folic acid or vitamin B12 deficiency, haemolytic anaemia, haemoglobinopathies, iron granulocytic anaemia, G6PD deficiency, etc.
6. Requirement for emergency surgical intervention.
7. Severe hepatic or renal impairment, ALT >3 times the upper limit of normal value or AST >3 times the upper limit of normal value, creatinine >1.5 times the upper limit of normal value
8. Pregnant or lactating women
9. history of blood transfusion, intravenous iron or ascorbic acid use within 12 weeks prior to surgery
10. Acute blood loss, gastrointestinal bleeding, etc. in the preoperative period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-04 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative allogeneic red blood cell transfusion volume | From the initiation of the surgical procedure until five days post-surgery.
  The volume of allogeneic red blood cell transfusions during the perioperative period.

SECONDARY OUTCOMES:
The quantity and percentage of allogeneic blood products utilized during the perioperative period. | From the initiation of the surgical procedure until until 90± 7 days following the surgical procedure.
  This encompasses blood components such as plasma and platelets, erythrocytes.
The alterations in perioperative haemoglobin levels. | From the point of randomisation until 90± 7 days following the surgical procedure.
  Haemoglobin levels were assessed at various time intervals.
The alterations in ferritin levels and TSAT during the perioperative period. | From the point of randomisation until 90± 7 days following the surgical procedure.
  Ferritin and Transferrin Saturation values were assessed at various time intervals.
The alterations in reticulocyte levels during the perioperative period. | From the point of randomisation until 90± 7 days following the surgical procedure.
  Reticulocyte levels were measured at various time intervals.
The score measuring the quality of life after surgery. | From the point of randomisation until 90± 7 days following the surgical procedure.
  The findings are presented based on the EQ VAS score (0-100), which reflects the overall self-assessed health status. A higher score indicates a better health status. Additionally, the results are reported using the EQ-5D-3L Effectiveness Index (EQ-5D-3L) values (5-15), where a lower EQ-5D-3L value signifies a better state of health.
Incidence of perioperative complication within 90 days after major cardiac surgery | From the point of randomisation until 90± 7 days following the surgical procedure.
  The potential postoperative complications within acute kidney injury (AKI), serious adverse events (SAE), congestive heart failure, respiratory failure, Allergic reaction, Thrombotic and thromboembolic complications and various infections.
The mortality rate within 30-day and 90-day postoperative period. | Within 90± 7 days after surgery
  The mortality rate within 30-day and 90-day postoperative period.
length of stay in hospital | Within 90± 7 days after surgery
  The time period from admission to the hospital to discharge
Length of stay in ICU | Within 90± 7 days after surgery
  The time period from admission to ICU after surgery to move out from ICU to normal ward

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Other researchers could email us to ask the data information.

REFERENCES:
- [Background] Zeroual N, Blin C, Saour M, David H, Aouinti S, Picot MC, Colson PH, Gaudard P. Restrictive Transfusion Strategy after Cardiac Surgery. Anesthesiology. 2021 Mar 1;134(3):370-380. doi: 10.1097/ALN.0000000000003682. PMID 33475735
- [Background] Fowler AJ, Ahmad T, Abbott TEF, Torrance HD, Wouters PF, De Hert S, Lobo SM, Rasmussen LS, Della Rocca G, Beattie WS, Wijeysundera DN, Pearse RM; International Surgical Outcomes Study Group. Association of preoperative anaemia with postoperative morbidity and mortality: an observational cohort study in low-, middle-, and high-income countries. Br J Anaesth. 2018 Dec;121(6):1227-1235. doi: 10.1016/j.bja.2018.08.026. Epub 2018 Oct 25. PMID 30442249
- [Background] Carson JL, Brittenham GM. How I treat anemia with red blood cell transfusion and iron. Blood. 2023 Aug 31;142(9):777-785. doi: 10.1182/blood.2022018521. PMID 36315909
- [Background] Spahn DR, Schoenrath F, Spahn GH, Seifert B, Stein P, Theusinger OM, Kaserer A, Hegemann I, Hofmann A, Maisano F, Falk V. Effect of ultra-short-term treatment of patients with iron deficiency or anaemia undergoing cardiac surgery: a prospective randomised trial. Lancet. 2019 Jun 1;393(10187):2201-2212. doi: 10.1016/S0140-6736(18)32555-8. Epub 2019 Apr 26. PMID 31036337
- [Background] Attallah N, Osman-Malik Y, Frinak S, Besarab A. Effect of intravenous ascorbic acid in hemodialysis patients with EPO-hyporesponsive anemia and hyperferritinemia. Am J Kidney Dis. 2006 Apr;47(4):644-54. doi: 10.1053/j.ajkd.2005.12.025. PMID 16564942